CLINICAL TRIAL: NCT02261077
Title: A Randomised, Double-blind, Placebo-controlled Study to Assess Pharmacokinetics, Safety and Tolerability of Single Rising Oral Doses (20 mg, 60 mg, 100 mg, 200 mg and 400 mg) and Multiple Rising Oral Doses (3 x 20 mg, 3 x 60 mg and 3 x 100 mg Per Day) of Buscopan® in Healthy Male Volunteers
Brief Title: Pharmacokinetics, Safety and Tolerability of Rising Doses of Buscopan® in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202.833
Record Dates: First submitted 2014-10-09; First posted 2014-10-10 (Estimated); Last update posted 2014-10-10 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
MeSH Terms: interventions — Butylscopolammonium Bromide

ARMS (3):
- Buscopan, single rising doses (Experimental)
  Interventions: Drug: Hyoscine butylbromide
- Buscopan, multiple rising doses (Experimental)
  Interventions: Drug: Hyoscine butylbromide
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hyoscine butylbromide
  Other Names: Buscopan®
  Arms: Buscopan, multiple rising doses; Buscopan, single rising doses
Drug: Placebo
  Arms: Placebo

SUMMARY:
Study to investigate pharmacokinetics, safety and tolerability of Buscopan® after single rising dose and after multiple rising doses

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males based upon a complete medical history, including the physical examination, vital signs (BP, PR), 12-lead ECG, clinical laboratory tests. There is no finding deviating from normal and of clinical relevance. There is no evidence of a clinically relevant concomitant disease.
2. Age ≥21 and age ≤50 years
3. BMI ≥18.5 and BMI <30 kg/m2 (Body Mass Index)
4. Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice and the local legislation

Exclusion Criteria:

1. Any finding of the medical examination (including BP, PR and ECG) deviating from normal and of clinical relevance
2. Evidence of a clinically relevant concomitant disease
3. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
4. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
5. History of relevant orthostatic hypotension, fainting spells or blackouts
6. Chronic or relevant acute infections
7. History of relevant allergy/hypersensitivity (including allergy to drug or its excipients) as judged clinically relevant by the investigator
8. Intake of drugs with a long half-life (> 24 hours) within at least one month or less than 10 half-lives of the respective drug prior to randomization
9. Use of drugs which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation within 10 days prior to enrolment in the study or during the study
10. Participation in another trial with an investigational drug within two months prior to randomization
11. Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
12. Inability to refrain from smoking on trial days as judged by the investigator
13. Alcohol abuse (more than 40 g/day for males)
14. Drug abuse
15. Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
16. Excessive physical activities within one week prior to administration or during the trial
17. Any laboratory value outside the reference range that is of clinical relevance
18. Inability to comply with dietary regimen of trial site
19. Hypersensitivity to hyoscine butylbromide and/or related drugs of these classes
20. History of megacolon
21. History of prostatic hyperplasia
22. History of mechanical stenosis of the gastrointestinal (e.g. after surgery of the gastrointestinal tract)
23. History of narrow-angle glaucoma
24. History of tachycardic arrhythmias
25. History of myasthenia gravis
26. Bladder-neck obstruction

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2007-05; Primary Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Maximum measured concentration of analyte in plasma (Cmax) | up to 104 hours after last drug administration
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) | up to 104 hours after last drug administration
Amount of analyte eliminated in urine from the time point t1 to time point t2 (Aet1-t2) | up to 80 hours after last drug administration

SECONDARY OUTCOMES:
Time from dosing to maximum measured concentration (tmax) | up to 104 hours after last drug administration
Area under the concentration-time curve of the analyte in plasma over a uniform dosing interval τ after administration of the first dose (AUCτ,1) | up to 32 hours after drug administration
Terminal rate constant in plasma (λz) | up to 104 hours after last drug administration
Terminal half-life of the analyte in plasma (t1/2) | up to 104 hours after last drug administration
Mean residence time of the analyte in the body (MRTpo) | up to 104 hours after last drug administration
Total/apparent clearance in plasma after extravascular administration (CL/F) | up to 104 hours after last drug administration
Apparent volume of distribution during the terminal phase λz following an extravascular dose (Vz/F) | up to 104 hours after last drug administration
Amount of analyte eliminated in urine from the time point t1 to time point t2 (Aet1-t2) | up to 80 hours after last drug administration
Fraction of analyte eliminated in urine from time point t1 to time point t2 (fet1-t2) | up to 80 hours after last drug administration
Renal clearance of the analyte from the time point t1 until the time point t2 (CLR,t1-t2) | up to 80 hours after last drug administration
Average concentration of the analyte in plasma at steady-state (Cavg) | up to 104 hours after last drug administration
Minimum concentration of the analyte in plasma at steady state over a uniform dosing interval τ (Cmin,ss) | up to 104 hours after last drug administration
Predose concentration of the analyte in plasma at steady state immediately before administration of the next dose (Cpre,ss) | predose on days 1-4
Linearity index (LI) | up to 104 hours after last drug administration
Accumulation ratio (RA) based on Cmax (RA,Cmax,N) | up to 104 hours after last drug administration
RA,AUC,N based on AUC0-τ | up to 104 hours after last drug administration
Number of subjects with clinically relevant findings in vital sign parameters (blood pressure (BP), pulse rate (PR)) | up to 14 days after last drug administration
Number of subjects with clinically relevant findings in 12-lead electrocardiogram | up to 14 days after last drug administration
Number of subjects with abnormal changes in laboratory parameters | up to 14 days after last drug administration
Number of subjects with abnormal findings in physical examination | up to 14 days after last drug administration
Occurrence of adverse events | up to 47 days
Tolerability assessed by investigator on a 4-point scale | within 14 days after last drug administration